CLINICAL TRIAL: NCT01410591
Title: The Effect of TIPS With 8- or 10-mm Covered Stent for Preventing Variceal Rebleeding in Cirrhotic Patients.
Brief Title: TIPS With 8- OR 10-mm Covered Stent for Preventing Variceal Rebleeding
Acronym: T8/10SVB
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Air Force Military Medical University, China (Other)
Responsible Party: Principal Investigator, Guohong Han, Head of Department of Digestive Interventional Radiology, Air Force Military Medical University, China
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: T8/10CSVB; FMMU-XHDD 003 (Registry Identifier: Fourth Military Medical University)
Record Dates: First submitted 2011-08-04; First posted 2011-08-05 (Estimated); Last update posted 2016-01-26 (Estimated); Status verified 2016-01

CONDITIONS: Decompensated Cirrhosis; Portal Hypertension; Bleeding Varices
Keywords: transjugular intrahepatic portosystemic shunt; TIPS; liver cirrhosis; variceal bleeding; 8- or 10-mm covered stent
MeSH Terms: conditions — Hypertension, Portal; Liver Cirrhosis

ARMS (2):
- 10-mm covered stent group (Active Comparator): Patients treated with 10-mm covered stent.
  Interventions: Device: 10-mm covered stent group
- 8-mm covered stent group (Active Comparator): Patients treated with 8-mm covered stent.
  Interventions: Device: 8-mm covered stent group

INTERVENTIONS:
Device: 8-mm covered stent group — Creating a shunt between hepatic vein and portal vein with a 8-mm covered stent by TIPS procedure.
  Arms: 8-mm covered stent group
Device: 10-mm covered stent group — Creating a shunt between hepatic vein and portal vein with a 10-mm covered stent by TIPS procedure.
  Arms: 10-mm covered stent group

SUMMARY:
The purpose of this study is to determine whether transjugular intrahepatic portosystemic shunt (TIPS) with 10-mm covered stent is associated with lower shunt dysfunction in comparing TIPS with 8-mm covered stent in cirrhotic patients with at least one episode of variceal bleeding.

ELIGIBILITY:
Inclusion Criteria:

* Cirrhotic patients with at least one episode of variceal bleeding
* No active bleeding within 5 days before TIPS
* Child-Pugh score ≤13
* Signed written informed consent

Exclusion Criteria:

* An age <18 years or >75 years
* With TIPS contraindications
* Past or present history of hepatic encephalopathy
* Pregnancy or breast-feeding
* Hepatic carcinoma and/or other malignancy diseases
* Sepsis
* Spontaneous bacterial peritonitis
* Uncontrollable hypertension
* Serious cardiac or pulmonary dysfunction
* Renal failure
* Portal vein thrombosis
* History of organ transplantation
* History of HIV (human immunodeficiency viruses) infection

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 127 (Actual)
Dates: Start 2012-07; Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Incidence of shunt dysfunction. | 2 years

SECONDARY OUTCOMES:
Incidence of variceal rebleeding | 2 years
Incidence of hepatic encephalopathy | 2 years
Survival | 2 years
Incidence of hepatic myelopathy | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Guohong Han, PhD & MD, Principal Investigator — Xijing Hospital of Digestive Diseases, Fourth Military Medical University
Locations (1):
- Xijing Hospital of Digestive Diseases, Fourth Military Medical University, Xi'an, Shaanxi, China

REFERENCES:
- [Background] Riggio O, Ridola L, Angeloni S, Cerini F, Pasquale C, Attili AF, Fanelli F, Merli M, Salvatori FM. Clinical efficacy of transjugular intrahepatic portosystemic shunt created with covered stents with different diameters: results of a randomized controlled trial. J Hepatol. 2010 Aug;53(2):267-72. doi: 10.1016/j.jhep.2010.02.033. Epub 2010 Apr 27. PMID 20537753
- [Derived] Wang Q, Lv Y, Bai M, Wang Z, Liu H, He C, Niu J, Guo W, Luo B, Yin Z, Bai W, Chen H, Wang E, Xia D, Li X, Yuan J, Han N, Cai H, Li T, Xie H, Xia J, Wang J, Zhang H, Wu K, Fan D, Han G. Eight millimetre covered TIPS does not compromise shunt function but reduces hepatic encephalopathy in preventing variceal rebleeding. J Hepatol. 2017 Sep;67(3):508-516. doi: 10.1016/j.jhep.2017.05.006. Epub 2017 May 12. PMID 28506905